CLINICAL TRIAL: NCT00384969
Title: A Phase I Study of Sorafenib and RAD001 in Patients With Metastatic Renal Cell Carcinoma
Brief Title: Sorafenib and RAD001 Renal Cell Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Charles Ryan, Clinical Professor of Medicine and Urology, University of California, San Francisco
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCSF06523
Record Dates: First submitted 2006-10-03; First posted 2006-10-06 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Renal Cell Carcinoma
Keywords: RAD001; Sorafenib; Renal Cell Carcinoma; Metastatic
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis | interventions — Everolimus; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): RAD001 and Sorafenib
  Interventions: Drug: RAD001 and Sorafenib

INTERVENTIONS:
Drug: RAD001 and Sorafenib — RAD001 2.5mg to 10.0mg PO QD Sorafenib 400mg PO BID

SUMMARY:
The objective of the phase I part of the study is to determine the maximum tolerated dose and dose limiting toxicities of the combination of RAD001 and sorafenib in patients with untreated metastatic kidney cancer.

DETAILED DESCRIPTION:
Phase I of the study will be an open-label dose escalation study to determine the MTD of the combination of sorafenib and RAD001. There will be a 7-day sorafenib run-in period prior to starting of RAD001 during cycle 1 to determine the pharmacokinetic effect of adding RAD001 on sorafenib drug levels. Starting doses will be set at RAD001 2.5 mg PO QD and sorafenib 400mg PO BID, continuously. Cycle length will be 4 weeks. Between 3 and 18 patients will be treated in the phase I portion of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically- or cytologically-confirmed renal cell carcinoma containing predominant (>50%) clear cell histology, which is metastatic or unresectable
2. Cytoreductive nephrectomy is allowed
3. Evidence of RECIST-defined measurable disease (lesions that can be accurately measured in at least one dimension with the longest diameter ≥ 20mm using conventional techniques or ≥10 mm with spiral CT scan)
4. Male or female at least 21 years old
5. ECOG performance status 0-1
6. Adequate bone marrow function:

   1. ANC ≥ 1500/uL
   2. platelet count ≥ 100,000/uL
   3. hemoglobin ≥ 9.0 g/dL
7. Adequate hepatic function:

   1. Total bilirubin ≤ 1.5 X ULN
   2. AST (SGOT) ≤ 2.5 X ULN
   3. ALT (SGPT) ≤ 2.5 X ULN
8. Adequate renal function as determined by either:

   1. Calculated or measured creatinine clearance ≥ 40 mL/min (for calculated creatinine clearance, Cockroft-Gault equation will be used) Modified Cockcroft-Gault formula: ((140 - age(yrs)) x (actual weight(kg))) / (72 x serum creatinine(mg/dl))

      * Multiply by another factor of 0.85 if female
   2. Serum creatinine ≤ 1.5 X ULN
9. Able to swallow oral medications
10. Resolution of any pre-existing toxicity from prior therapy to NCI CTCAE V3.0 ≤ grade 1
11. Signed and dated informed consent document
12. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures
13. More than 28 days since any prior therapy, including investigational agents and surgical procedures

Exclusion Criteria:

1. Collecting duct, papillary, or chromophobe type renal cell carcinoma without a clear cell component are excluded. Transitional cell carcinoma of the renal pelvis is excluded
2. No more than two prior systemic regimens for renal cell carcinoma
3. Phase I: No prior treatment with sorafenib. Phase II: No prior treatment with prior anti-VEGF therapies, including sorafenib, sunitinib, thalidomide, or bevacizumab
4. No prior treatment with RAD001, CCI-779, or similar agents
5. Prior surgery, radiation therapy, or systemic therapy for renal cell carcinoma within 4 weeks of starting study treatment
6. History of or known brain metastasis, spinal cord compression, or carcinomatous meningitis, or new evidence of brain or leptomeningeal disease on screening CT or MRI scan
7. Any of the following within 12 months prior to study drug administration: myocardial infarction, unstable or severe angina, coronary or peripheral artery bypass graft, NYHA functional Class II, III, IV congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism
8. Hypertension that is unable to be controlled with medications
9. Known human immunodeficiency virus (HIV) or acquired immune deficiency syndrome (AIDS)-related illness
10. "Currently active" second malignancy other than non-melanoma skin cancers. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are considered to have a less than 30% risk of relapse
11. Current treatment on another clinical trial
12. Pregnant or breastfeeding
13. Chronic treatment with systemic steroids or other immunosuppressive agent
14. Patients with an active bleeding diathesis or on oral vitamin K antagonist medication (except low dose warfarin)
15. History of malabsorption syndrome, disease significantly affecting gastrointestinal function or major resection of stomach or small bowel that could interfere with absorption, distribution, metabolism, or excretion of study drugs
16. Any serious and/or unstable pre-existing medical, psychiatric, or other condition (including lab abnormalities) that could interfere with subject safety or obtaining informed consent. Examples of such include uncontrolled diabetes, nonhealing wound, severe infection, severe malnutrition, ventricular arrhythmias, active ischemic heart disease, chronic liver or renal disease, or active upper GI tract ulceration -

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2006-10; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | weekly

SECONDARY OUTCOMES:
Objective response rate | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Charles Ryan, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States